CLINICAL TRIAL: NCT04522908
Title: A Phase II Study Evaluating Reduced Starting Dose and Dose Escalation of Cabozantinib as Second-line Therapy for Advanced HCC in Patients With Preserved Liver Function
Brief Title: Dose Escalation Study of Cabozantinib for Advanced HCC Patients With Preserved Liver Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Johann Wolfgang Goethe University Hospital, Prof. Dr. med. Trojan (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CaboRISE; 2020-000775-20 (EudraCT Number); AIO-HEP-0320/ass (Other: Arbeitsgemeinschaft Internistische Onkologie)
Record Dates: First submitted 2020-08-03; First posted 2020-08-21 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma (HCC); Second Line Treatment
Keywords: hepatocellular carcinoma; HCC; Child-Pugh A
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — cabozantinib

STUDY DESIGN:
Intervention Model Description: Clinical trials with a single arm, all eligible patients will receive Cabozantinib starting dose of 40 mg, oral, once daily for 4 weeks, followed by Cabozantinib escalated dose of 60 mg, oral, once daily from week 5 onwards
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cabozantinib - Single Arm (Experimental): Single Arm with Cabozantinib starting dose 40 mg for 4 weeks and dose escalation to 60 mg afterwards.
  Interventions: Drug: Cabozantinib Oral Tablet

INTERVENTIONS:
Drug: Cabozantinib Oral Tablet — Cabozantinib starting dose of 40 mg, oral, once daily for 4 weeks followed by Cabozantinib escalated dose of 60 mg, oral, once daily from week 5 onwards
  Other Names: CABOMETYX

SUMMARY:
Open-label, single arm, multicenter phase II trial assessing the tolerability of a reduced starting dose of 40 mg cabozantinib for 4 weeks and subsequent dose escalation to 60 mg cabozantinib until disease progression or intolerable toxicities.

DETAILED DESCRIPTION:
The primary objective is to assess the tolerability of a reduced starting dose of 40 mg cabozantinib once-daily for 4 weeks and subsequent dose escalation to 60 mg cabozantinib once-daily to be maintained until disease progression or intolerable toxicities. Using the same study treatment discontinuation criteria as in the pivotal CELESTIAL trial will allow for comparison of treatment discontinuation rates due to treatment related adverse events (TRAEs) defined as unresolved intolerable Grade 2 TRAEs or any unresolved Grade 3 TRAEs (see Section 6).

Patients eligible for this trial are HCC patients with preserved liver function previously treated with any first line therapy.

Secondary objectives comprise the assessment of overall survival (OS), progression free survival (PFS) at 10 weeks, objective response rate (ORR), time on treatment, treatment exposure (dose intensity/dose reductions), toxicity, and quality of life (QLQ-C30).

In addition, tissue samples (optional) will be analyzed for molecular parameters and immune cell composition to identify biomarkers potentially associated with clinical efficacy (OS, PFS and ORR).

This is an open label, single-arm, multicenter phase II trial. 40 patients suffering from advanced stage hepatocellular carcinoma (HCC) with preserved liver function in second line treatment, after any first line therapy, will be enrolled in this trial.

Patients will be recruited from up to 10 sites and patients withdrawn from the trial will not be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Fully-informed written consent.
* Males and females ≥ 18 years of age.

  *There are no data that indicate special gender distribution. Therefore, patients will be enrolled in the study gender-independently.
* Patients with HCC who have been previously treated with any first line therapy.
* Locally advanced or metastatic and/or unresectable HCC with preserved liver function (Child-Pugh A only, if liver cirrhosis is present) with diagnosis confirmed by histology/cytology or clinically by guideline criteria.
* Disease that is not amenable to curative surgical and/or locoregional therapies, or progressive disease after surgical and/or locoregional therapies.
* ECOG performance status ≤ 2.
* Resolution of any acute, clinically significant treatment-related toxicity from prior therapy to Grade 1 prior to study entry, with the exception of alopecia.
* Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.
* For women of childbearing potential (WOCBP): agreement to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive methods from the time of signing the informed consent through at least 4 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse. Male patients, even if surgically sterilized (i.e. status post-vasectomy) must agree to practice effective barrier contraception (e.g. condom) and to refrain from sperm donation during the entire study treatment period and through at least 4 months after the last dose of study drug or agree to completely abstain from heterosexual intercourse.

Exclusion Criteria:

* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within at least 4 months.
* Significant portal hypertension (moderate or severe ascites). Significant hypertension, defined as blood pressure ≥ 140 mmHg (systolic) or ≥ 90 mmHg (diastolic) in repeated measurements.
* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* Patients with impaired liver function defined as Child-Pugh B or C, if liver cirrhosis is present.
* Severely impaired kidney function (defined as creatinine > 2 mg/dl and/or creatinine clearance < 45 mL/min).
* Elevations of AST/ALT > 5 x ULN at baseline.
* Presence of encephalopathy in past 12 months.
* Significant cardiovascular disease (such as NYHA Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina.
* Baseline QTcF > 500 ms.
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study.
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
* Treatment with investigational systemic therapy within 28 days or five times the elimination half-life of the investigational product, whichever is longer, prior to initiation of study treatment.
* Prior cabozantinib use.
* Known or suspected hypersensitivity to cabozantinib or any other excipients of the IMP.
* Rare hereditary galactose intolerance, total lactase deficiency or glucose-galactose malabsorption.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.
* Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Treatment discontinuation rate due to treatment-related adverse events | 27 months
  Any unresolved intolerable Grade 2 TRAE or unresolved Grade ≥ 3 TRAE after 60 mg or 40 mg or any intolerable Grade 2 TRAE or Grade ≥ 3 TRAE after 20 mg will count as treatment discontinuation due to AE.

SECONDARY OUTCOMES:
Overall survival | 27 months
  Time from the date of enrollment to the date of death from any cause. Subjects who have not died by the date of data cutoff will be right censored at the last known date alive.
Progression free survival (PFS) according to RECIST 1.1 | at 10 weeks
  Time from the date of enrollment to the date of first observed disease progression (investigator assessment according to RECIST 1.1) or death from any cause. Subjects who have died without a reported disease progression will be considered to have progressed on the date of their death. Subjects who did not progress or have died will be right censored on the date of their last evaluable tumor assessment.
Objective response rate (ORR) according to RECIST 1.1 | 27 months
  Objective response rate will be assessed according to RECIST 1.1 (refer to Appendix 5). Objective response rate will be defined as the proportion of subjects experiencing a confirmed complete response (CR) or confirmed partial response (PR) per RECIST 1.1.
Time on treatment | 27 months
  Time on treatment defined as the interval from therapy initiation until premature discontinuation.
Treatment exposure | 27 months
  Treatment exposure defined as summary of specific dose intensities on treatment (including dose reductions and interruptions).
Treatment-related and -unrelated toxicities (AEs, SAEs) according to NCI CTCAE v5.0 | 27 months
  All observed treatment-related and -unrelated toxicities (type, incidence and severity of AEs and SAEs) and side effects will be graded according to NCI CTCAE v5.0 and the degree of association of each with the study treatment assessed and summarized. The treatment related serious adverse events rate (SAE) will be determined.
Quality of Life with the EORTC QLQ-C30 patient questionnaire | 27 months
  Patient reported outcome assessed by the validated EORTC patient quality of life questionnaire QLQ-C30. The questionnaire evaluates the patient's health and activities in everyday life. Values reach from 1 (not at all) to 4 (very much). Low values mean a better outcome.
Correlation of biomarkers potentially associated with clinical efficacy (OS, PFS and ORR) | 27 months
  The TR projects might include the assessment of the following:
  FFPE tissue for IHC staining; FFPE tissue for nucleic isolation to assess the expression of biomarkers, determination of genetic alterations in HCC (panel sequencing) or to determine the mutational load.

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Chair — Frankfurter Institut fuer Klinische Krebsforschung IKF GmbH
Locations (10):
- Germany (10):
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Universitätsklinikum Köln AöR, Cologne
  - BAG / Onkologische Gemeinschaftspraxis, Dresden
  - Ev. Kliniken Essen-Mitte, Klinik für Internistische Onkologie, Essen
  - Universitätsklinikum Essen, Essen
  - Institute for Clinical Cancer Research Krankenhaus Nordwest, Frankfurt
  - Klinikum der Johann-Wolfgang-Goethe Universität, Frankfurt
  - Universitätsklinikum Gießen und Marburg, Giessen
  - Universität Leipzig KöR, Medizinische Fakultät Department für Innere Medizin, Neurologie Klinik für Gastroenterologie, Leipzig
  - Klinikum rechts der Isar Technische Universität München Klinik und Poliklinik für Innere Medizin II, Müchen

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared